CLINICAL TRIAL: NCT05817513
Title: Effect of Myofascial Release on Spinal Curvature, Pre Menstrual Symptoms and Quality of Life in Scoliotic Females With Dysmenorrhea.
Brief Title: Effect of Myofascial Release on Scoliotic Females With Dysmenorrhea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Liza ibrahim saadallah ibrahim, Liza Ibrahim saadallah ibrahim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 012/004351
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Scoliosis Idiopathic Adolescent; Dysmenorrhea; Premenstrual Syndrome; Quality of Life
Keywords: Scoliosis , dysmenorrhea, Myofascial release, pre Menstrual symptoms
MeSH Terms: conditions — Dysmenorrhea; Premenstrual Syndrome; Scoliosis | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Two groups, one group will be treated by traditional exercises for scoliosis treatment and another group will be treated by Myofascial release and traditional exercises.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): (Control group): will consist of 26 young females . They will receive traditional exercises for scoliosis.
  Interventions: Other: Traditional exercises for scoliosis treatment.
- (Study group) (Experimental): (Study group): will consist of 26 young females. They will receive the same traditional scoliosis exercises in addition to myofascial release ( MFR ) .
  Interventions: Other: Myofascial release.; Other: Traditional exercises for scoliosis treatment.

INTERVENTIONS:
Other: Myofascial release. — Myofascial release (MFR) is a therapeutic treatment that uses gentle pressure and stretching to facilitate the release of fascial restrictions caused by accidents, injury, stress, repetitive use, and traumatic or surgical scarring. The fascial restrictions are palpated by the practitioner and the techniques are applied directly to the skin of the patient without lotions or oils. The pressure is applied into the direction of the restriction just until resistance is felt or the tissue is perceived to stop moving. The pressure is sustained at this point of resistance, without sliding over the skin or forcing the tissue, for a minimum of 90-120s. As the tissue begins to release, the practitioner maintains the same amount of pressure and follows the release three dimensionally through multiple releases.
  Arms: (Study group)
Other: Traditional exercises for scoliosis treatment. — The exercises are:
  1. Pelvic tilt.
  2. Arm and leg raises.
  3. Cat-cow.
  4. Bird dog.
  5. Latismus dorsi stretch.
  6. Abdominal press.
  7. Practice a good posture.
  8. Stretching and scapular exercises.

SUMMARY:
PURPOSE:

The purpose of this study is to determine the effect of myofascial release on spinal curvature, premenstrual symptoms, and quality of life in scoliotic females with dysmenorrhea

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a complex 3D structural disorder of the spine seen in children from 10 years old until skeletal maturity and confirmed by a Cobb angle of 10° or more and accompanied by vertebral rotation (Addai et al., 2020). It is the most common types of scoliosis and it is predominantly seen in girls at low curve magnitudes ( LeBauer et al., 2008).

A previous study reported the beneficial effect of myofascial release (MFR) on adults with idiopathic scoliosis (LeBauer et al., 2008). MFR showed a decrease in pain, improved posture, and advancement in quality of life, which may include physical, social, and pulmonary function (las Penas, 2005). HYPOTHESES:

There will be no effect of myofascial release on spinal curvatures, menstrual pain, and quality of life in young scoliotic females with primary dysmenorrhea .

ELIGIBILITY:
Inclusion Criteria:

1. All young females have primary dysmenorrhea and idiopathic scoliosis.
2. They are diagnosed with idiopathic scoliosis; their trunk rotation and rib hump measured by scoliometer will be more than 5.
3. They will experience pain in abdominal region, back and/or referred to the thigh during menstruation.
4. They experience a regular menstrual cycle
5. Their age will range from 18 to 25 years old.
6. Body mass index (BMI) will range between 18.5 to 24.9 kg/m2.

Exclusion Criteria:

1. Females who have any pelvic diseases or secondary dysmenorrhea.
2. Females who had received any spinal surgeries.
3. Females with irregular menstrual cycles.
4. History of gynecological interventions and having received manipulative treatment within the 2 months before the beginning of the study.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of trunk rotation and rib hump by Scoliometer. | Eight weeks.
  Scoliometer will be used to measure trunk rotation and rib hump of each female in both groups (A&B) at starting and after the end of the treatment course. The most common method to screen for significant scoliosis is the forward bend test, which is often combined with the use of a sociometer

SECONDARY OUTCOMES:
Premenstrual symptoms were assessed using MSQ questionnaire. | Eight weeks.
  Premenstrual symptoms were assessed using MSQ questionnaire a modified version of MOO's.
  The symptoms commonly found are assessed on a four point scale with response ranging from 0 =no effect; 1 = mild, present; 2 = moderate; and 3 = severe disabling with regard to It evaluated behavioral changes; water and salt retention; depression. The MSQ also measured the occurrence and severity of two menstrual pain symptoms including cramp and backache experienced during the first 2 days of the subjects' last menstrual period.
Assessment of quality of life by ISYQOL QUESTIONNAIRE (Italian Spine Youth Quality of Life (ISYQOL) Measuring Spine Related Quality of Life) | Eight weeks.
  ISYQOL QUESTIONNAIRE(Italian Spine Youth Quality of Life (ISYQOL) Measuring Spine Related Quality of Life):The Italian Spine Youth Quality of Life questionnaire (ISYQOL) measures the health-related quality of life of adolescents with spinal deformities.ISYQOL consists of 20 items, each scored 0, 1 or 2. In accordance with the Rasch analysis technique, used to develop the questionnaire, the ordinal ISYQOL total score is converted to an interval measure (i.e., ISYQOL measure), which is expressed on a 0%- 100% scale (with 100% indicating high quality of life). Seven ISYQOL items assess the impact of bracing on quality of life and these are to be administered only to individuals who actually wear a brace. Thanks to the Rasch analysis approach, it is possible to compare the ISYQOL result of non-brace wearers (who answer only 13 of the 20 items) with that of brace wearers (who complete the entire questionnaire).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No